CLINICAL TRIAL: NCT03743233
Title: Hand and Engine-driven Techniques for Endodontic Retreatment: Randomized Clinical Trial
Brief Title: Hand and Engine-driven Techniques for Endodontic Retreatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PPGO027
Record Dates: First submitted 2018-10-16; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand file instrumentation (Active Comparator)
  Interventions: Device: Reciprocating
- Reciprocating instrumentation (Active Comparator)
  Interventions: Device: Hand file

INTERVENTIONS:
Device: Hand file — A crown-down technique will be performed until reaching the provisory WL. The root canals will be initially deobstructed with size #3 and #2 Gates-Glidden burs (Dentsply-Maillefer) at the coronal and middle root thirds. Then, hand stainless steel K-files (Dentsply-Maillefer) with decreasing sizes will be used (#40, #35, #30, #25). The WL will be determined by an electronic apex locator (Novapex; Forum Technologies, Rishon Le-Zion, Israel). A radiograph will be taken to confirm the WL, which should be 1 mm short of the root apex. Apical patency will be reached and maintained with a size #15 K-file (Dentsply-Maillefer). The root canals will be reinstrumented and a size #50 K-file will be standardized as the master apical instrument. A step-back procedure in 1-mm increments followed until merging with the crown-down rotary enlargement (size #70) will be achieved.
  Arms: Reciprocating instrumentation
Device: Reciprocating — Reciproc R25 file will be used for gutta-percha removal, until reaching the WL. The instrument will be introduced into the canal applying slight movements of 3-mm amplitude. Apical patency will be maintained with a size #15 K-file. The root canals will be reinstrumented using the Reciproc R50 file. For both groups, after the root canal filling removal and reinstrumentation protocol, a new radiograph will be taken, without any intracanal instrument, for posterior analysis of the percentage of remaining filling material in the root canal. If the radiograph demonstrates the persistence of filling material, the technique will be repeated with the last instrument used in the chemomechanical preparation (hand or reciprocating file), also using H-files with circumferential movements against the dentinal walls in order to remove these residual material, followed by abundant irrigation with NaOCl.
  Arms: Hand file instrumentation

SUMMARY:
Numerous instrumentation techniques have been suggested for the nonsurgical retreatment of teeth with primary failure of endodontic therapy in laboratory studies. However, there is limited clinical evidence about those different techniques. The objective of this study is to compare the prevalence and intensity of postoperative pain, as well as the success rate after endodontic retreatment with hand or engine-driven reciprocating instrumentation. A randomized clinical trial will be performed, considering two comparison groups: hand preparation with stainless steel instruments or engine-driven reciprocating preparation with the Reciproc NiTi System (VDW, Munich, Germany), to verify which technique would lead to lower postoperative pain levels and higher endodontic success rates. Secondary outcomes related to technique efficiency will be also registered, evaluating the capacity of filling material removal and the time spent on the clinical procedures. Eighty individuals who need endodontic retreatment in single-rooted teeth will be selected (n=40/group). Endodontic reintervention will be carried out in two visits. Periapical radiographs taken after root filling removal protocols will be transferred to an image analysis software. Then, the percentage of remaining filling material in relation to the total area of the root canal will be evaluated. The clinical time spent with the removal procedure protocol will be registered, in minutes, by a digital stopwatch. After each visit, postoperative pain will be assessed using a numerical rating scale. The record of pain and analgesic drug intake will be performed in 12, 24, 48 hours and 7 days after the clinical procedures. Success rates will be evaluated after 3, 6, 12 and 24 months, through clinical and radiographic examination, considering the Periapical Index, a 5-point score system. Data of both groups (percentage of remaining debris, operating time, postoperative pain, clinical and radiographic success) will be analyzed for normality by the Shapiro-Wilk test. Assuming normal distribution, the data will be compared by t test. Pearson's correlation coefficient will be applied to detect possible correlations between the evaluated outcomes. Differences will be considered significant at P=0.05.

ELIGIBILITY:
Inclusion Criteria:

* Good systemic and oral health;
* Requiring root canal retreatment in single-rooted teeth (one root and one root canal);
* Asymptomatic persistent apical periodontitis.

Exclusion Criteria:

* Use of analgesics, anti-inflammatory drugs or other pain modulating drugs;
* Chronic systemic disease (eg: diabetes, hypertension, arthritis and renal dysfunction);
* Systemic disease that could interfere with bone quality;
* Pregnant or breastfeeding women;
* Teeth with untreated periodontal disease;
* Abnormal mobility and with excessively large or curved canals.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Post operative pain | 12, 24, 48 hours and 7 days
  Change of post operative pain from baseline to 12h, from 12 to 24h, from 24 to 48h and from 48h to 7 days after treatment, assessed using a visual analog scale, where "zero" means no pain and "10" means maximum pain possible

SECONDARY OUTCOMES:
Periapical index | Radiographs will be taken after 3, 6, 12 and 24 months
  the radiograph will be assessed considering the apex of the tooth and changes occurred after 3, 6, 12 and 24months after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No